CLINICAL TRIAL: NCT04176211
Title: The Impact of Myasthenia Gravis in the Real World
Status: Completed | Type: Observational
Sponsor: Vitaccess Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 5105-08-2019
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis Disease; Neuromuscular Diseases; Neuromuscular Junction Diseases; Nervous System Diseases; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Ocular Myasthenia Gravis; Generalized Myasthenia Gravis; Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis; Neuromuscular Diseases; Neuromuscular Junction Diseases; Nervous System Diseases; Autoimmune Diseases; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An international, non-interventional, prospective, community recruited, longitudinal, lifestyle study which aims to collect Real-World Evidence (RWE) from people living with myasthenia gravis (MG) in order to map the disease's natural history, its burden on patients and their families, its treatment, as well as its medical, social and pharmacoeconomic impact.

DETAILED DESCRIPTION:
Data was collected from people with MG using the MyRealWorld™ RWE platform , developed by the healthcare digital research company, Vitaccess. Participants downloaded a 'bring your own device' (BYOD) study app, MyRealWorld™ MG, onto their smartphones, which they used to enter data and complete surveys about their MG.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years and over) with any stage and any subtype of myasthenia gravis disease
* Resident in Belgium, Canada, France, Germany, Italy, Japan, Spain, the UK, the USA, or Denmark

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age >18 years) with any stage and any subtype of myasthenia gravis disease
Sampling Method: Non-Probability Sample
Enrollment: 2847 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in EuroQol 5-dimension 5-level (EQ-5D-5L) score | Monthly throughout 2 year study duration
  The EQ-5D-5L comprises two parts - the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (EQ VAS).
  The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems - i.e., higher scores represent worse health). The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
  The EQ VAS records the respondent's self-rated health on vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. Higher scores represent better self-perceived health.
Change in Myasthenia Gravis Activities of Daily Living (MG-ADL) score | Four times per six months throughout 2 year study duration
  The MG-ADL is a myasthenia gravis-specific 8-item scale, which assesses the severity of the following symptoms: talking, chewing, swallowing, breathing, impairment of ability to brush teeth/comb hair, impairment of ability to rise from a chair, double vision, and eyelid droop. Each of the 8 items has 4 response options; 0 (Mild), 1 (Moderate), 2 (Mild) and 3 (Severe). The MG-ADL total score can be calculated by totalling all 8 items out of a maximum score of 24. A higher score indicates severe impairment.
Change in Myasthenia Gravis Quality of Life 15-item revised scale (MG-QoL15r) score | Once per six months throughout 2 year study duration
  The MG-QOL15r is a myasthenia gravis-specific health-related quality of life survey, which assesses the impact of myasthenia gravis over the past few weeks on the following domains: emotions, physical health, self-care, social life, and impact on role. Each of the 15 items has three response options: 0 (Not at all), 1 (Somewhat), and 2 (Very much). The MG-QoL15r total score can be calculated by totalling all 15 items out a maximum score of 30. A higher score indicates severe impairment.
Change in Hospital Anxiety and Depression Scale (HADS) score | Once per six months throughout 2 year study duration
  The HADS is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. It consists of two subscales, Anxiety and Depression. The instrument comprises 14 items, 7 for the anxiety subscale and 7 for the depression subscale. Each item is scored on a 4-point response scale, scale wording changes for each item with each coding response corresponding with greater impairment or severity. Domain scores can be calculated by totalling all 7 items out of a maximum score of 21. High scores indicate greater severity of that impairment
Change in Health Utilities Index III (HUI3) score | Once per 12 months throughout 2 year study duration
  The HUI3 is a generic 8-item survey, which provides descriptive evidence on multiple dimensions of health status, a score for each dimension of health, and a health-related quality of life score for overall health.Health dimensions include vision, hearing, speech, ambulation/mobility, pain, dexterity, emotion and cognition. Each dimension has five or six response options. It has recall periods of either 'usual health', the past week, two weeks, or four weeks. Scores on individual items are combined to given a combined health state which can then be converted to health utilities. Lower health utilities represent worse health.
COVID-19 survey results | Monthly throughout 2 year study duration
  This is a bespoke survey designed to understand the impact of COVID-19 on study participants. It includes questions about whether participants have had COVID, and the consequences if so, whether they have been vaccinated, and how the wider pandemic has affected their MG treatment and quality of life.
Change in Single Simple Question (SSQ) and Patient Acceptable Symptom States (PASS) scores | Four times per six months throughout 2 year study duration
  The SSQ is a single question that asks respondents what percentage of normal they feel with respect to their MG. The PASS is a single question that asks respondents whether they would consider their current disease state to be satisfactory if they had to stay in it for the next few months. The SSQ and PASS will be presented to participants at the same time, as a question pair.
Change in EuroQol 5-dimension 3-level (EQ-5D-3L) score | Monthly for three months for participants from the US and Italy only
  The EQ-5D-3L is a three-level version of the EQ-5D-5L. It includes the same dimensions as the EQ-5D-5L, but each has only three levels: no problems, some problems, and extreme problems. The EQ VAS is unchanged from the EQ-5D-5L version.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Dyspnea Characteristics score | Once per six months throughout 2 year study duration
  The PROMIS sleep disturbance measure assesses self-reported frequency, severity, and duration of dyspnea (shortness of breath) over the last 7 days using either a 0-10 numeric rating scale or 0-4 rating scale to assess dyspnea characteristics.Each item is evaluated individually according to the numeric rating scale. No total score is calculated for this instrument. Higher scores on items indicate more severe symptoms.
Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score | Once per six months throughout 2 year study duration
  The FACIT-Fatigue measure is a generic 13-item survey which assesses fatigue levels and impact over the past 7 days. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigue to 0 = very much fatigued). Scores range from 0-52. The higher the score, the better the quality of life.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance short form 6a change | Once per six months throughout 2 year study duration
  The PROMIS sleep disturbance measure assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep over the last 7 days using a 5-point scale. Scores range from 6-30. Higher scores represent worse sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Mark JW Larkin, PhD, Principal Investigator — Vitaccess Ltd
Locations (1):
- Vitaccess Ltd, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated data may be available via application.

REFERENCES:
- [Background] Berrih-Aknin S, Claeys KG, Law N, Mantegazza R, Murai H, Sacca F, Dewilde S, Janssen MF, Bagshaw E, Kousoulakou H, Larkin M, Beauchamp J, Leighton T, Paci S. Patient-reportedimpact of myasthenia gravis in the real world: protocol for a digital observational study (MyRealWorld MG). BMJ Open. 2021 Jul 20;11(7):e048198. doi: 10.1136/bmjopen-2020-048198. PMID 34285010
- [Result] Dewilde S, Philips G, Paci S, Beauchamp J, Chiroli S, Quinn C, Day L, Larkin M, Palace J, Berrih-Aknin S, Claeys KG, Muppidi S, Mantegazza R, Sacca F, Meisel A, Bassez G, Murai H, Janssen MF. Patient-reported burden of myasthenia gravis: baseline results of the international prospective, observational, longitudinal real-world digital study MyRealWorld-MG. BMJ Open. 2023 Jan 31;13(1):e066445. doi: 10.1136/bmjopen-2022-066445. PMID 36720569
- [Result] Berrih-Aknin S, Palace J, Meisel A, Claeys KG, Muppidi S, Sacca F, Amini F, Larkin M, Quinn C, Beauchamp J, Philips G, De Ruyck F, Ramirez J, Paci S. Patient-reported impact of myasthenia gravis in the real world: findings from a digital observational survey-based study (MyRealWorld MG). BMJ Open. 2023 May 11;13(5):e068104. doi: 10.1136/bmjopen-2022-068104. PMID 37169499
- [Derived] Janssen MF, Dewilde S, Wolfe GI, Muppidi S, Phillips G. Psychometric properties of MG-ADL items and MG-ADL score: An assessment of distributional characteristics, validity and factor structure in two large datasets. J Neurol Sci. 2024 Aug 15;463:123135. doi: 10.1016/j.jns.2024.123135. Epub 2024 Jul 22. PMID 39068745